CLINICAL TRIAL: NCT00385658
Title: A 16-week Multicenter, 2-period Study to Investigate the Effect of the Combination of Fluvastatin ER 80mg and Fenofibrate 200mg on HDL-C in Comparison to the Combination of Simvastatin 20mg and Ezetimibe 10mg in Patients With Metabolic Syndrome
Brief Title: Efficacy of Fluvastatin and Fenofibrate in Comparison to Simvastatin and Ezetimibe in Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CXUO320BDE35
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia; metabolic syndrome; fluvastatin; fenofibrate; simvastatin; ezetimibe
MeSH Terms: conditions — Dyslipidemias; Metabolic Syndrome | interventions — Fenofibrate; Ezetimibe

INTERVENTIONS:
Drug: Fluvastatin extended release, fenofibrate
Drug: Fixed combination simvastatin/ezetimibe

SUMMARY:
This study will investigate the effects of the combination of fluvastatin and fenofibrate on dyslipidemia in comparison to the combination of simvastatin and ezetimibe.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study prior to any study procedures.
* Male or female subjects, age between 18-75 years inclusive.
* All women of child bearing potential must have a negative pregnancy test
* Metabolic Syndrome according to the International Diabetes Federation definition:

  * Low plasma HDL-C (Men < 40 mg/dl ; Women < 50 mg/dl ).
  * Elevated waist circumference (men ≥ 94 cm, women ≥ 80cm)
  * And one or more of the following criteria:

    * Triglycerides ≥ 150 mg/d.l
    * Raised blood pressure (DBP ≥ 85 mmHg and/or SBP ≥ 130mmHg ) or treated hypertension.
    * Fasting plasma glucose≥ 100mg/dl.
    * Previously diagnosed type 2 diabetes.

Exclusion Criteria:

* Dyslipidemia secondary to other causes such as nephrotic syndrome, autoimmune disease.
* Type 1 diabetes.
* HbA1c > 9.5%.
* Unexplained serum creatine phosphokinase > 2 x Upper limit of normal.
* History of myocardial infarction and/or cerebral stroke and/or unstable angina pectoris.
* Known or suspected contraindications and warnings according to the country specific label for the investigational drugs.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
High density lipoprotein cholesterol (HDL-C) measured at the end of each study period.

SECONDARY OUTCOMES:
Compared at the end of each treatment period:
patients reaching target levels of low density lipoprotein cholesterol (LDL-C) <100mg/dl
patients reaching target levels of non-HDL-C <130mg/
LDL-C/HDL-C
Triglycerides
LDL subfractions in a subgroup of patients

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Director — Novartis
Locations (2):
- Investigative Centers, Germany
- Novartis Pharma AG, Basel, Switzerland